CLINICAL TRIAL: NCT00604344
Title: A 48-week, Randomised, Multi-centre, Openlabelled, Parallel-group Trial to Compare the Efficacy and the Safety of NN304 (Insulin Detemir) and NPH Human Insulin in Subjects With Insulin Requiring Diabetes Mellitus on a Basal-bolus Regimen
Brief Title: Efficacy and the Safety of Insulin Detemir in Subjects With Insulin Requiring Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1476; JapicCTI-R070008 (Registry Identifier: JAPIC)
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin NPH

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to investigate the efficacy of insulin detemir on blood glucose control in subjects with insulin requiring diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Duration of diabetes mellitus for at least 2 years
* Current treatment of basal-bolus regimen for at least 12 weeks using an intermediate/long-acting human insulin and insulin aspart
* HbA1C below 11.0%

Exclusion Criteria:

* Impaired renal function
* Impaired hepatic function
* Serious heart diseases
* Known hypoglycaemia unawareness or recurrent major hypoglycaemia
* Proliferative retinopathy or maculopathy requiring acute treatment
* Uncontrolled treated/untreated hypertension
* Current treatment with total insulin dose of more than 100 IU/day
* Current treatment or expected at the screening to start treatment with systemic corticosteroids

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2003-04; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 48 weeks of treatment

SECONDARY OUTCOMES:
Blood glucose profiles
Hypoglycaemic episodes
Adverse events
Body weight
Insulin antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Kobayashi M, Iwamoto Y, Kaku K, Kawamori R, Tajima N. 48-week Randomized Multicenter Open-label Parallel Group Phase 3 Trial to Compare Insulin Detemir and NPH Insulin Efficacy and Safety in Subjects with Insulin Requriring Diabetes Mellitus in a Basal-bolus Regimen. J. Japan Diab. Soc 2007; 50 (9): 649-663
- [Result] Kobayashi M, Iwamoto Y, Kawamori R, Tajima N, Nishida T, Kaku K. Insulin detemir achieves lower, less variable fasting glucose and a reduced risk of nocturnal hypoglycaemia and weight gain compared to NPH insulin in basal bolus therapy of Japanese patients with type 1 diabetes. Diabetologia 2006; 49 (Suppl 1): A608-A609 [Abstract 995]
- [Result] Ishii H, Iwamoto Y, Kaku K, Kawamori R, Tajima N, Kobayashi M. Quality of Life (QoL) Assessment of Insulin Detemir and NPH Human Insulin in Japanese Subjects with Diabetes on Basal-Bolus Regimen. Diabetes 2007; 56 (Suppl. 1): A170 (2805-PO)
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com